CLINICAL TRIAL: NCT04913129
Title: The Burden of COVID-19 Survivorship: Exercise Therapy to Combat the Sequelae of COVID-19
Brief Title: The Burden of COVID-19 Survivorship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan Taylor, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-002693
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard physician-guided medical care after COVID-19
- Interventional (exercise training) Group (Experimental): 8 week home-based exercise training
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — 8 week home-based exercise therapy 4-5 times/week
  Arms: Interventional (exercise training) Group

SUMMARY:
This research study is being done to find out what the longer-term physiological consequences of COVID-19 are, and to determine if exercise therapy can help improve lung function, heart function and overall fitness, and reduce symptoms in people recovering from SARS-CoV-2.

DETAILED DESCRIPTION:
The purpose of this research is to see if taking part in structured exercise training will improve the ability to exercise, the function of the lungs and the function of the heart, and reduce symptoms of fatigue and breathlessness in people recovering from COVID-19. After enrollment all patients will complete exercise testing, lung function testing, and cardiac imaging. Patients will be randomized to either 8 weeks of exercise training (4-5 times per week) or will continue standard medical care. All patients will undergo detailed exercise testing, lung function testing, and cardiac imaging after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 75 years.
* History of RT-PCR proven SARS-CoV-2 infection.
* Deemed 'recovered' from SARS-CoV-2 infection.
* Not clinically obese (BMI ≥ 36) and/or suffer from musculoskeletal or other conditions that would limit exercise participation.
* No evidence of cardiac ischemia at rest or during exertion (via ECG).
* Able to provide written informed consent.

Exclusion Criteria:

* Individuals less than 21 or more than 75 years old.
* Not able to take part in structured exercise training due to injury or other conditions that would put person at risk during exercise.
* Unable to provide written informed consent.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen update (VO2max) measured in mL/kg/min | 8 weeks
  VO2max is the maximal oxygen consumed during an exhaustive exercise test

SECONDARY OUTCOMES:
Peak exercise work rate (Wpeak) measured in Watts | 8 weeks
  Wpeak is the highest achieved power during a maximal incremental cycle exercise test
Forced vital capacity (FVC) measured in L | 8 weeks
  FVC is the largest amount of air that can be exhaled from the lungs in one maximal breath
Forced expiratory volume in 1 second (FEV1) measured in L | 8 weeks
  FEV1 is the largest amount of air that can be exhaled from the lungs in the first second of one maximal breath
Maximal inspiratory pressure (MIP) measured in cmH2O | 8 weeks
  Highest inspiratory muscle pressure (i.e. inspiratory muscle strength) during a maximal inspiratory effort
Maximal expiratory pressure (MEP) measured in cmH2O | 8 weeks
  Highest expiratory muscle pressure (i.e. expiratory muscle strength) during a maximal expiratory effort
Left ventricular contractile function measured as % fractional area change (LV FAC) | 8 weeks
  LV FAC is a measure of overall contractile function of the LV
Right ventricular contractile function measured as % fractional area change (RV FAC) | 8 weeks
  RV FAC is a measure of overall contractile function of the RV

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Taylor, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials